CLINICAL TRIAL: NCT05926232
Title: Expanded Access for Repotrectinib
Status: Available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA127-1057
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

MeSH Terms: interventions — repotrectinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Repotrectinib — Repotrectinib
  Other Names: BMS-986472

SUMMARY:
This is an expanded access designed to provide access to Repotrectinib for eligible participants.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Pre-Approval Access (PAA) Healthcare Practitioner Requests — https://www.bms.com/healthcare-providers/early-patient-access-to-investigational-medicine/investigational-drugs-available.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm